CLINICAL TRIAL: NCT02447783
Title: Effect of Cocoa Flavanol Intake on Blood Pressure and Platelet Function in Healthy Adults, Part 2
Brief Title: Effect of Long Term Cocoa Flavanol Intake on Blood Pressure and Platelet Function in Healthy Adults, Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 311497-II; 311497-II (Other: UC Davis)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Flavanols; Cocoa flavanols; Blood pressure; Platelet Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control, Flavanol-free intervention (Placebo Comparator): Intake of flavanol-free, macro- and micro-nutrient matched control capsules
  Interventions: Dietary Supplement: Control Capsules
- CF intervention (Active Comparator): Intake of capsules containing Mars Cocoa Extract Capsules manufactured by the Cocoapro® process and providing 500 mg of cocoa flavanols per capsule
  Interventions: Dietary Supplement: Mars Cocoa Extract Capsules

INTERVENTIONS:
Dietary Supplement: Control Capsules — Cocoa-based, flavanol-free, control-matched capsules consumed for 12 weeks (Week 1: 2 capsules/day; Week 2: 3 capsules/day; Week 3-12: 4 capsules/day; Week 12-14: no capsule intake).
  Arms: Control, Flavanol-free intervention
Dietary Supplement: Mars Cocoa Extract Capsules — Capsules containing Mars Cocoa Extract manufactured by the Cocoapro® process and containing 500 mg of cocoa flavanols per capsule consumed for 12 weeks (Week 1: 2 capsules/day; Week 2: 3 capsules/day; Week 3-12: 4 capsules/day; Week 12-14: no capsule intake).
  Arms: CF intervention

SUMMARY:
Flavanols are plant-derived compounds commonly present in the human diet. Examples of flavanol-containing foods and beverages are apples, chocolate, tea, wine, berries, pomegranate and nuts. The consumption of flavanol-containing foods and beverages has been associated with improvements in cardiovascular health. In this study, the investigators hope to learn more about the effects of long term consumptions of cocoa flavanols on blood pressure, platelet function and other metabolic parameters in healthy humans. This study is a continuation of a previous study investigating the consumptions of increasing amounts of cocoa flavanols on blood pressure, platelet function and other metabolic parameters in healthy humans

ELIGIBILITY:
Inclusion Criteria:

* 30-55 years old
* A normal blood chemistry and liver function
* BMI < 30 kg/m2
* previously consumed cocoa and peanut products, with no adverse reactions

Exclusion Criteria:

* A history of cardiovascular disease, stroke, hypertension, renal, hepatic, or thyroid disease, GI tract disorders, previous GI surgery, metabolic syndrome, diabetes, taking cholesterol-lowering medication, hormone replacement therapy, antioxidant supplements, on aspirin therapy or taking anticoagulants, or on a medically prescribed diet.
* Allergies to nuts, cocoa and chocolate products
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, on a weight loss diet or using herbal dietary supplements

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline (day 0) and 6,12 and 14 weeks after intervention
  Blood pressure will be measured using standard techniques.

SECONDARY OUTCOMES:
Change in platelet function | Baseline and 6, 12 and 14 weeks after intervention
  Platelet function will be determined using the PFA-100® analyzer (Dade Behring International, Miami, FL) with collagen-epinephrine (CEPI)- and collagen-ADP (CADP) stimulation.
Change in 24 h ambulatory blood pressure | Baseline (day 0) and 12 weeks after intervention
  24 h ambulatory blood pressure will be measured using standard techniques.
Change in metabolic parameters in blood | Baseline (day 0) and 6, 12 and 14 weeks after intervention
  Metabolic parameters determined in blood included: comprehensive metabolic panel, liver panel and cell blood counting.

OTHER OUTCOMES:
Change in plasma concentration of cocoa flavanol metabolites | Baseline (day 0) and 6, 12 and 14 weeks after intervention
  Cocoa flavanol metabolites in plasma include: structurally related (-)-epicatechin metabolites and 5-(3,4-dihydroxyphenyl)-4-valerolactone metabolites
Change in plasma concentration of methylxanthines | Baseline (day 0) and 6, 12, and 14 weeks after intervention
  Methylxanthines determined in plasma include: caffeine, theobromine, paraxanthine and theophylline

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — UC Davis
Locations (1):
- Ragle Human Nutrition Research Center, Department of Nutrition at UC Davis, Davis, California, United States

REFERENCES:
- [Background] Schroeter H, Heiss C, Spencer JP, Keen CL, Lupton JR, Schmitz HH. Recommending flavanols and procyanidins for cardiovascular health: current knowledge and future needs. Mol Aspects Med. 2010 Dec;31(6):546-57. doi: 10.1016/j.mam.2010.09.008. Epub 2010 Sep 18. PMID 20854838
- [Derived] Ottaviani JI, Balz M, Kimball J, Ensunsa JL, Fong R, Momma TY, Kwik-Uribe C, Schroeter H, Keen CL. Safety and efficacy of cocoa flavanol intake in healthy adults: a randomized, controlled, double-masked trial. Am J Clin Nutr. 2015 Dec;102(6):1425-35. doi: 10.3945/ajcn.115.116178. Epub 2015 Nov 4. PMID 26537937